CLINICAL TRIAL: NCT04345315
Title: Correlative Study on Cancer Patients and Healthcare Professionals Exposed to SARS-CoV-2 Infection
Brief Title: Correlative Study on Cancer Patients and Healthcare Professionals Exposed to Infection by Severe Acute Respiratory Syndrome-Corona Virus-2 (SARS-Cov-2), COVID-19 Causative Agent.
Acronym: CORSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: AUSL Romagna (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRSTB113
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: SARS-CoV-2; COVID-19; cancer; IgM-IgG; seroprevalence
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — Serologic Tests; High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — oropharyngeal and nasal swabs and blood samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- asymptomatic population at high risk of infection: healthy individuals at high risk of infection, including individuals who have had contact with a patient tested positive for COVID-19, voluntary health workers and oncological patients candidate to immunosuppressive therapy
  Interventions: Other: serological test; Other: Rapid molecular test; Other: serum chemistry analysis
- COVID-19 patients: patients with confirmed diagnosis of COVID-19
  Interventions: Genetic: Next generation Sequencing (NGS) analysis

INTERVENTIONS:
Other: serological test — serological test assessing IgM and IgG directed against SARS-CoV-2
  Groups: asymptomatic population at high risk of infection
Other: Rapid molecular test — Molecular test to detect SARS-CoV-2 in oro/rhinopharyngeal swab
  Groups: asymptomatic population at high risk of infection
Genetic: Next generation Sequencing (NGS) analysis — analysis of genetic variability of virus and host
  Groups: COVID-19 patients
Other: serum chemistry analysis — Analysis of serum chemistry factors and coagulation panel in blood samples
  Groups: asymptomatic population at high risk of infection

SUMMARY:
Translational, prospective / retrospective, non-profit, non-pharmacological study, with cohort characteristics.

The study consists of two parts: the first to study epidemiological aspects of the spread of the disease and the second one to identify infection-related genetic factors.

DETAILED DESCRIPTION:
The outbreak of COVID-19 infections is spreading in Italy with unprecedented severity characteristics. In this context, it is essential to collect data relating to the epidemiology of the disease, to outline further useful tools for diagnosis and to define the correct use of rapid molecular and / or serological tests in the surveillance of high-risk subjects (cancer patients and healthcare operators), in order to identify any new disease control strategies, crucial to reduce the transmission and to outline specific guidelines for cancer patients healthcare management. It is also necessary to identify the factors that determine the evolution of the viral genome over time in the various geographical areas and also the potential susceptibility markers in the different types of affected subjects (symptomatic, mildly symptomatic and asymptomatic).

ELIGIBILITY:
For epidemiologic analysis:

Inclusion Criteria:

* Age > 18 years
* asymptomatic
* One of the following three conditions: • Healthy subjects who have had contact with COVID-19 positive patients • Healthcare workers • oncological patients candidates for cytotoxic chemotherapy at myeloablative doses (such as transplants) or treated with immune-check point inhibitors.
* informed consent to the study and processing of data

Exclusion Criteria:

* presence of symptoms for COronaVIrus Disease 19 (COVID-19) (fever > 37.5 °, cough, shortness of breath)

For analysis of viral/host genetic factors involved in susceptibility/resistance to infection, samples from patients with confirmed diagnosis of COVID-19, residual from diagnostic procedures will be analyzed. All samples for genetic analysis will be anonymized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For epidemiologic analysis, asymptomatic population 350 health workers / healthy subjects at risk of infection and 50 cancer patients candidates for immunosuppressive therapies will be enrolled.
  For analysis of genetic variability of virus and host factors impacting on susceptibility to infection: samples from about 100 SARS-CoV-2 positive patients (sintomatic, paucisintomatic or asymptomatic), retained at Pievesestina Laboratory after diagnostic procedure, will be analyzed. All samples for genetic analysis will be anonymized.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
epidemiology | 12 months
  Investigate the epidemiology of the infection in an asymptomatic population including both healthy individuals at high risk of infection and oncological patients by assessing the seroprevalence of IgG and IgM antibodies against the SARS-CoV-2

SECONDARY OUTCOMES:
Immunoglobulin G (IgG) and Immunoglobulin M (IgM) antibodies evaluation | 12 months
  IgG and IgM antibodies evaluation over time
methods comparison | 24 months
  Make a comparison between different serological investigation methods and rapid molecular methods becoming available
correlation between biochemical and coagulative factors with SARS-CoV-2 positivity. | 24 months
  To evaluate correlation between biochemical and coagulative factors with SARS-CoV-2 positivity
phylogenetic map | 24 months
  Building a phylogenetic map of an epidemic Italian macro-region
interactions between the virus and host cells | 24 months
  Evaluate the spectrum of possible interactions between the virus and host cells, considering their genetic variability / instability in patients diagnosed with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Prof., Principal Investigator — IRST IRCCS
Locations (2):
- Italy (2):
  - UO Microbiologia,Centro Servizi Pievesestina, AUSL Romagna, Cesena, FC
  - Irst Irccs, Meldola, FC

IPD SHARING:
Plan to Share IPD: No